CLINICAL TRIAL: NCT00234793
Title: Maternal Problem-Solving in Childhood Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, OJ Sahler, Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: RO1 CA098964-02; RSRB 09840
Record Dates: First submitted 2005-09-12; First posted 2005-10-07 (Estimated); Last update posted 2015-06-15 (Estimated); Status verified 2015-06

CONDITIONS: Stress; Cancer
Keywords: childhood cancer; intervention; maternal coping; problem solving skills; anxiety; cope; problem solving
MeSH Terms: conditions — Neoplasms; Anxiety Disorders

INTERVENTIONS:
Behavioral: Problem-Solving Skills Training

SUMMARY:
The purpose of this study is to help mothers of children with cancer to cope more effectively by increasing their problem-solving skills.

DETAILED DESCRIPTION:
The purpose of this study is:

1. to develop a time-and-attention control condition to better assess the direct and mediational effect of PSST independent of social support (placebo);
2. to develop a personal digital assistant hand-held supplement to standard PSST to provide real-time training, reinforcement, and on-the-spot documentation of PSST usage;
3. to develop independent measures of the application of problem-solving strategies in everyday life; and
4. to measure utilization of and satisfaction with other resources accessed by mothers as independent indicators of the usefulness and cost-effectiveness of PSST.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of any age with a child diagnosed with any form of cancer 2-16 weeks prior to contact.

Exclusion Criteria:

* Mothers of children with cancer if they do not read or speak English or Spanish, if their child is in severe medical crisis, or if they live a prohibitive distance to complete the intervention.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2003-05; Study Completion 2010-04

PRIMARY OUTCOMES:
The primary aim of the study is to evaluate the effectiveness of problem-solving training provided to mothers of children with newly diagnosed cancer in decreasing negative affectivity
e.g. depression, anxiety, and increasing satisfaction with resource utilization

SECONDARY OUTCOMES:
Standardized measures at three time points: pre-intervention, post-intervention, 3 months post the second time point

CONTACTS AND LOCATIONS:
Overall Officials: Olle Jane Z. Sahler, MD, Principal Investigator — University of Rochester; Robert W Butler, PhD, Principal Investigator — Oregon Health and Science University; Martha A Askins, PhD, Principal Investigator — M.D. Anderson Cancer Center; Robert B Noll, PhD, Principal Investigator — University of Pittsburgh; Ernest R Katz, PhD, Principal Investigator — Children's Hospital Los Angeles; Donna R Copeland, PhD, Principal Investigator — UT/MD Anderson Cancer Center; Lewis W Johnson, PhD, Study Director — University of Southern California
Locations (4):
- United States (4):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Oregon Health Sciences University, Portland, Oregon
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - UT/MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Result] Askins MA, Sahler OJ, Sherman SA, Fairclough DL, Butler RW, Katz ER, Dolgin MJ, Varni JW, Noll RB, Phipps S. Report from a multi-institutional randomized clinical trial examining computer-assisted problem-solving skills training for English- and Spanish-speaking mothers of children with newly diagnosed cancer. J Pediatr Psychol. 2009 Jun;34(5):551-63. doi: 10.1093/jpepsy/jsn124. Epub 2008 Dec 17. PMID 19091804
- [Derived] Sahler OJ, Dolgin MJ, Phipps S, Fairclough DL, Askins MA, Katz ER, Noll RB, Butler RW. Specificity of problem-solving skills training in mothers of children newly diagnosed with cancer: results of a multisite randomized clinical trial. J Clin Oncol. 2013 Apr 1;31(10):1329-35. doi: 10.1200/JCO.2011.39.1870. Epub 2013 Jan 28. PMID 23358975